CLINICAL TRIAL: NCT03141814
Title: A Better Understanding of Molecular Mechanisms Leading to Asthma and Its Remission
Brief Title: Asthma Origins and Remission Study
Acronym: ARMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Maarten van den Berge, MD PhD, University Medical Center Groningen
Other Study IDs: NL2015001
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sputum bronchial biopsies bronchial brushes nasal brushes particles in exhaled air
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- asthma: 20 patients with ongoing ashma
- complete asthma remission: 20 subjects with complete asthma remission
- clinical asthma remission: 20 subjects with clinical asthma remission
- non-asthmatic healthy controls: 20 subjects without respiratory symptoms and normal lung function and no bronchial hyperresponsiveness to methacholine and/or AMP

SUMMARY:
Asthma is characterized by chronic airway inflammation of the large and small airways. Asthma patients often have episodes with symptoms of dyspnea, wheezing and nocturnal awakening. Currently available inhaled anti-inflammatory treatments reduce the airway inflammation and treatment but do not cure the disease. Therefore asthma patients often need life-long treatment to control their asthma.

In a small subset of patients, their asthma resolves spontaneously. This phenomenon is called asthma remission. Subjects with asthma remission do not experience symptoms or signs of airway inflammation anymore and do not require inhaled treatments. Some subjects with asthma remission also have a completely normal lung function without signs of bronchial hyperresponsivess: they have complete asthma remission. Unfortunately, asthma remission occurs only in a small subset of 15-25% of asthma patients.Objective: to determine the underlying mechanisms and molecular events leading to remission of asthma.

DETAILED DESCRIPTION:
Rationale: Asthma inception occurs only in susceptible individuals, and is often triggered by specific environmental factors, such as respiratory viruses and aeroallergens. Although asthma is generally viewed as a chronic persistent disease, remission of asthma is possible in a subset of patients. This is highly relevant, since understanding mechanisms that contribute to asthma inception and remission may teach us how asthma can be stopped and thus may provide novel avenues for the treatment of asthma. In adulthood, average remission rates of asthma are approximate 2% per year 1. We observed that remission in adulthood is more likely with earlier onset of asthma, less airway obstruction, more severe bronchial hyperresponsiveness, and smoking cessation. A proper definition of remission is very important; we therefore introduced the terms 'clinical remission' and 'complete remission' 2. Clinical remission was defined as the absence of asthma symptoms and no use of asthma medication, complete remission as the absence of asthma symptoms, no use of asthma medication, normal lung function and no bronchial hyperresponsiveness. In a longitudinal study of 119 allergic asthmatic children followed-up for 30 years, our group found that clinical remission occurred in 30% and complete remission in 22% of all cases.

Objective: to determine the underlying mechanisms and molecular events involved in the inception and remission of asthma.

Methods: We will include a 40 subjects divided over the following 4 groups: i) clinical asthma remission (10 subjects), ii) complete asthma remission (10 subjects), iii) ongoing asthma (10 patients), iv) non-asthmatic healthy controls (10 subjects) in a cross-sectional study. All subjects will be extensively clinically characterized including respiratory symptoms/questionnaires, in- and expiratory CT-scans, and parameters of large and small airway function and inflammation. In addition, blood and nasal epithelial brushes will be obtained to study the genetic and epigenetic mechanisms of asthma remission. Finally, bronchoscopy with bronchial biopsies and brushes will be performed under conscious sedation. Bronchial biopsies from all four patient groups will be used for index FACS sorting of the three most important cell types orchestrating the asthmatic inflammatory process: i.e. B lymphocytes, CD4+ T cells and CD8+ T cells. We will perform single cell whole-genome transcriptome sequencing on at least 100 cells of each type and the primary outcome of the study is to identify how the transcriptomic profile of bronchial epithelial cells is changed between asthma patients and healthy controls as a consequence of asthma inception and what transcriptomic profile changes occur in CD4+ CD8+ and B lymphocytes in the airways from subjects with asthma remission compared to patients with ongoing asthma and healthy controls.

ELIGIBILITY:
Inclusion criteria for all subjects:

* Age between 40 and 65 years old.
* Smoking history ≤ 10 packyears.

Inclusion criteria for all asthmatics and asthma remission subjects:

• Development of asthma symptoms before 21 years.

Specific inclusion criteria for the 4 different groups:

* Group 1. Subjects with clinical asthma remission:

  * Documented history of asthma diagnosed according to latest GINA guidelines, i.e. respiratory symptoms and either bronchodilator reversibility (improvement in FEV1 of more than 12% of baseline (and at least 200 mL) after inhalation of 800 µg salbutamol.
  * No use of asthma medications such as inhaled or oral corticosteroids, β2-agonists or anticholinergic in the last 3 years.
  * No symptoms of wheeze or asthma attacks during the last 3 years.
* Group 2. Subjects with complete asthma remission

  * Documented history of asthma diagnosed according to latest GINA guidelines, i.e. respiratory symptoms and either bronchodilator reversibility (improvement in FEV1 of more than 12% of baseline (and at least 200 mL) after inhalation of 800 µg salbutamol.
  * No use of asthma medications such as inhaled or oral corticosteroids, β2-agonists or anticholinergics in the last 3 years.
  * No symptoms of wheeze or asthma attacks during the last 3 years.
  * FEV1 > 90% predicted.
  * Absence of bronchial hyperresponsiveness, i.e. both PC20 methacholine > 8 mg/ml and PC20 AMP > 320 mg/ml.
* Group 3. Patients with ongoing asthma

  * Documented history of asthma diagnosed according to latest GINA guidelines, i.e. respiratory symptoms and either bronchodilator reversibility (improvement in FEV1 of more than 12% of baseline (and at least 200 mL) after inhalation of 800 µg salbutamol.
  * Use of inhaled corticosteroids or either persistent symptoms of wheeze, cough, or dyspnea or regular use of β2 agonists at least once a week during the last 2 months.
  * PC20 methacholine < 8 mg/ml.
* Group 4. Non-asthmatic controls

  * No history of asthma.
  * No use of inhaled corticosteroids or β2-agonists for a period longer than 1 month.
  * No symptoms of wheeze, nocturnal dyspnea, or bronchial hyperresponsiveness.
  * PC20 methacholine > 8 mg/ml, FEV1/FVC > 70% and FEV1 > 80% predicted.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * 20 patients with a documented history of asthma who have clinical asthma remission.
  * 20 patients with a documented history of asthma who have complete asthma remission.
  * 20 patients with current asthma.
  * 20 healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Single cell sequencing data | baseline
  Single cell mRNA sequencing of lymphocytes in bronchial biopsies and blood eosinophils

SECONDARY OUTCOMES:
Spirometry | baseline
  FEV1, FVC, FEV1/FVC, FEF25-75.
body box | baseline
  RV, RV/TLC, FRC, IC, ERV
HRCT | baseline
  emphysema and small airways disease
Airway inflammation | baseline
  Sputum, blood, biopsy inflammatory cell counts, exhaled nitric oxide, small particles in exhaled breath
Small airways disease | baseline
  Multiple breath nitrogen washout: LCI, Sacin, Scond
genetic and genome-wide mRNA, non-coding RNA, and DNA methylation | baseline
  assessed in bronchial and nasal epithelial brushes, biopsies and blood

CONTACTS AND LOCATIONS:
Overall Officials: Maarten van den Berge, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Netherlands